CLINICAL TRIAL: NCT01632488
Title: Assessment of Small Intestinal Bowel Epithelial Gaps in Patients With Irritable Bowel Syndrome by Confocal Laser Endomicroscopy
Brief Title: Assessment of Small Intestinal Bowel Epithelial Gaps in Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: 2012SDU-QILU-G02
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Disease
Keywords: Irritable Bowel Syndrome; Inflammatory Bowel Disease; Confocal Laser Endomicroscopy
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Taken biopsies during endoscopy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Irritable bowel syndrome: Patients admitted to outpatient department with symptoms meeting Rome III criteria of irritable bowel syndrome.
- Inflammation: Patients with long standing history or short onset of inflammatory bowel disease.
- Normal controls: Asymptomatic individuals admitted for health surveillance or patients for follow up after polypectomy.

SUMMARY:
The study aims to:

1. Determine whether the density of epithelial gaps in terminal ileum of patients with irritable bowel syndrome (IBS) is different from that in inflammatory bowel disease (IBD) patients and normal controls by confocal laser endomicroscopy (CLE).
2. Evaluate the relationship between the density of epithelial gaps and IBS subtypes, and visceral hypersensitivity.

DETAILED DESCRIPTION:
Epithelial cells lining the gastrointestinal tract serve as a barrier between the gut lumen and the body. Previous study has shown that epithelium is punctuated by discontinuities named "gaps". Confocal laser endomicroscopy could be used as a useful tool for detecting epithelial gaps in vivo, and epithelial gap density in terminal ileum of IBD patients was elevated compared with normal control using CLE. So this study aims to determine whether the density of epithelial gaps in terminal ileum of patients with IBS is different from that in IBD patients and normal controls by CLE, and to evaluate the relationship between the density of epithelial gaps and IBS subtypes, and visceral hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Bowel habits alterations meeting IBS Rome III criteria and indications for colonoscopy investigation
* Patients with history of inflammatory bowel disease
* Asymptomatic individuals for health surveillance or patients for follow up after polypectomy
* Patients complained of hemafecia but colonoscopy revealed only haemorrhoid

Exclusion Criteria:

* Patients with known cancers or abdominal surgery
* Alarm symptoms such as anaemia, gastrointestinal bleeding or obstruction, marked weight loss, abdominal mass
* Patients who are unwilling to sign or give the informed consent form
* Patients who are allergic to fluorescein sodium
* Patients with impaired cardiac, liver or renal function
* Patients with coagulopathy
* Patients with pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for colonoscopy in Qilu Hospital outpatient and inpatient department.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Facility: Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China